CLINICAL TRIAL: NCT01657162
Title: An Extension Study to Evaluate 24 Months of Standard-of-Care Osteoporosis Management Following Completion of 18 Months of BA058 or Placebo Treatment in Protocol BA058-05-003
Brief Title: Twenty-Four Month Extension Study of BA058-05-003 (Abaloparatide) in Participants With Osteoporosis
Acronym: ACTIVExtend
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA058-05-005; ACTIVExtend Trial (Other: Radius Health, Inc.); 2012-002216-10 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-06 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Postmenopausal Osteoporosis
Keywords: BA058; Abaloparatide-SC; abaloparatide; ACTIVExtend; osteoporosis; fracture; bone loss
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Fractures, Bone; Bone Diseases, Metabolic | interventions — Alendronate

STUDY DESIGN:
Masking Description: Even though this is an open-label study, participants and Investigators who will be participating in this study (BA058-05-005) will remain blinded to the prior treatment assignment in Study BA058-05-003 (NCT02653417) until all participants completed the first 6 months of BA058-05-005 for prespecified data analysis. Complete data analysis for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alendronate (Experimental): Participants received 70 milligrams (mg) of alendronate orally once per week beginning on Day 2 for up to 24 months after participating in Study BA058-05-003 during which participants received abaloparatide 80 micrograms (mcg) SC or abaloparatide-matching placebo daily for 18 months.
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — Alendronate is a bisphosphonate drug that prevents bone resorption by osteoclast and is used for the treatment of osteoporosis.
  Other Names: Fosamax; Alendronate sodium

SUMMARY:
The purpose of this study is to provide 24 months of standard of care data on participants previously enrolled in Study BA058-05-003 (NCT02653417).

DETAILED DESCRIPTION:
To assess the long-term effect of the anabolic drug, abaloparatide-subcutaneous (SC) versus placebo in the prevention of bone fracture after cessation of treatment. Participants who completed the 18-month Double-Blind BA058-05-003 (ACTIVE) study (NCT02653417), after receiving abaloparatide-SC or placebo, were enrolled in this extension study to receive 70 mg of alendronate (bisphosphonate) weekly for an additional 24 months. Complete details for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.

ELIGIBILITY:
Inclusion Criteria:

1. The participant was enrolled, randomized to either the abaloparatide-SC (BA058) or placebo arm, and successfully completed Study BA058-05-003 (NCT02653417).
2. The participant was no more than 40 days from End-of-Treatment (Month 18) in Study BA058-05-003 (NCT02653417).

Exclusion Criteria:

1. Participants who were withdrawn from Study BA058-05-003 (NCT02653417) for any reason.
2. Participants who experienced a treatment-related serious adverse event (SAE) during Study BA058-05-003 (NCT02653417).

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2012-11-20 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2016-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Mitlak, Study Director — Radius Health, Inc.
Locations (25):
- United States (3):
  - Lakewood, Colorado
  - Hialeah, Florida
  - Bethesda, Maryland
- Buenos Aires, Argentina
- Brazil (5):
  - Brasília
  - Curitiba
  - Rio de Janeiro
  - São Paulo
  - Vitória
- Czechia (3):
  - Brno
  - Brno-Vinohrady
  - Pardubice
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- Estonia (2):
  - Tallinn
  - Tartu
- Hong Kong, Hong Kong
- Vilnius, Lithuania
- Poland (5):
  - Bialystok
  - Kielce
  - Lodz
  - Warsaw
  - Zgierz
- Bucharest, Romania

REFERENCES:
- [Result] Cosman F, Miller PD, Williams GC, Hattersley G, Hu MY, Valter I, Fitzpatrick LA, Riis BJ, Christiansen C, Bilezikian JP, Black D. Eighteen Months of Treatment With Subcutaneous Abaloparatide Followed by 6 Months of Treatment With Alendronate in Postmenopausal Women With Osteoporosis: Results of the ACTIVExtend Trial. Mayo Clin Proc. 2017 Feb;92(2):200-210. doi: 10.1016/j.mayocp.2016.10.009. PMID 28160873
- [Result] Bone HG, Cosman F, Miller PD, Williams GC, Hattersley G, Hu MY, Fitzpatrick LA, Mitlak B, Papapoulos S, Rizzoli R, Dore RK, Bilezikian JP, Saag KG. ACTIVExtend: 24 Months of Alendronate After 18 Months of Abaloparatide or Placebo for Postmenopausal Osteoporosis. J Clin Endocrinol Metab. 2018 Aug 1;103(8):2949-2957. doi: 10.1210/jc.2018-00163. PMID 29800372
- [Derived] Cosman F, Hans D, Shevroja E, Wang Y, Mitlak B. Effect of Abaloparatide on Bone Microarchitecture Assessed by Trabecular Bone Score in Women With Osteoporosis: Post Hoc Analysis of ACTIVE and ACTIVExtend. J Bone Miner Res. 2023 Apr;38(4):464-470. doi: 10.1002/jbmr.4764. Epub 2023 Feb 12. PMID 36588166
- [Derived] Watts NB, Dore RK, Baim S, Mitlak B, Hattersley G, Wang Y, Rozental TD, LeBoff MS. Forearm bone mineral density and fracture incidence in postmenopausal women with osteoporosis: results from the ACTIVExtend phase 3 trial. Osteoporos Int. 2021 Jan;32(1):55-61. doi: 10.1007/s00198-020-05555-1. Epub 2020 Sep 15. PMID 32935170
- [Derived] Greenspan SL, Fitzpatrick LA, Mitlak B, Wang Y, Harvey NC, Deal C, Cosman F, McClung M. Abaloparatide followed by alendronate in women >/=80 years with osteoporosis: post hoc analysis of ACTIVExtend. Menopause. 2020 Oct;27(10):1137-1142. doi: 10.1097/GME.0000000000001593. PMID 32665529
- [Derived] Cosman F, Peterson LR, Towler DA, Mitlak B, Wang Y, Cummings SR. Cardiovascular Safety of Abaloparatide in Postmenopausal Women With Osteoporosis: Analysis From the ACTIVE Phase 3 Trial. J Clin Endocrinol Metab. 2020 Nov 1;105(11):3384-95. doi: 10.1210/clinem/dgaa450. PMID 32658264
- [Derived] Leder BZ, Mitlak B, Hu MY, Hattersley G, Bockman RS. Effect of Abaloparatide vs Alendronate on Fracture Risk Reduction in Postmenopausal Women With Osteoporosis. J Clin Endocrinol Metab. 2020 Mar 1;105(3):938-43. doi: 10.1210/clinem/dgz162. PMID 31674644
- [Derived] Leder BZ, Zapalowski C, Hu MY, Hattersley G, Lane NE, Singer AJ, Dore RK. Fracture and Bone Mineral Density Response by Baseline Risk in Patients Treated With Abaloparatide Followed by Alendronate: Results From the Phase 3 ACTIVExtend Trial. J Bone Miner Res. 2019 Dec;34(12):2213-2219. doi: 10.1002/jbmr.3848. Epub 2019 Sep 11. PMID 31411768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants who received abaloparatide or placebo in the double-blind study (BA058-05-003 [Study 003]), were enrolled to this open-label extension study. Complete results for Study 003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Pre-assignment Details: The procedures performed for the Follow-up visit (Month 19) for Study 003 served as Baseline for Day 1 of Study BA058-05-005 (Study 005).
Groups:
- Abaloparatide-SC/Alendronate: Participants received 70 milligrams (mg) of alendronate orally once per week beginning on Day 2 for up to 24 months after participating in Study BA058-05-003 during which participants received abaloparatide 80 micrograms (mcg) subcutaneous (SC) daily for 18 months.
- Placebo/Alendronate: Participants received 70 mg of alendronate orally once per week beginning on Day 2 for up to 24 months after participating in Study BA058-05-003 during which participants received abaloparatide-matching placebo daily for 18 months.
Period: Overall Study
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Started (Participants who started Study BA058-05-005.) | 558 | 581
Study 003 ITT Population (This Intent-To-Treat (ITT) population included participants who were randomized into Study 003.) | 824 (Participants received 80 mcg abaloparatide SC during Study 003.) | 821 (Participants received abaloparatide-matching placebo during Study 003.)
Study 003 Modified ITT (mITT) Population (Study003 ITT participants with Study 003 pretreatment & postbaseline evaluable radiologic assessment) | 690 (Participants received 80 mcg abaloparatide SC during Study 003.) | 711 (Participants received abaloparatide-matching placebo during Study 003.)
Completed Study 003 | 606 (Participants received 80 mcg abaloparatide SC during Study 003.) | 637 (Participants received abaloparatide-matching placebo during Study 003.)
Study 005 ITT Population (All Study 003 ITT participants who enrolled in Study 005 .) | 558 | 581
Study 005 Safety Population (All Study 005 ITT participants who received 1 or more doses of alendronate.) | 553 | 580
Study 005 mITT Population (Study 003 mITT participants with a Study 005 postbaseline evaluable radiologic test (spine X-ray)) | 544 | 568
Completed | 499 | 506
Not Completed | 59 | 75
Not completed — Adverse Event | 26 | 36
Not completed — Withdrawal by Subject | 13 | 13
Not completed — Continuing Significant Deterioration | 9 | 3
Not completed — Refusal of Treatment | 4 | 6
Not completed — Lost to Follow-up | 3 | 4
Not completed — Death | 2 | 3
Not completed — Inability to Complete Study Procedures | 1 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Hypersensitivity to Alendronate | 0 | 1
Not completed — Other than Specified | 0 | 2

BASELINE CHARACTERISTICS:
Population: Study BA058-05-005 ITT Population: all Study BA058-05-003 ITT participants who enrolled in the BA058-05-005 study. Study BA058-05-003 ITT population included all participants who were randomized into the BA058-05-003 study. Baseline Characteristics for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Groups:
- Abaloparatide-SC/Alendronate: Participants received 70 mg of alendronate orally once per week beginning on Day 2 for up to 24 months after participating in Study BA058-05-003 during which participants received abaloparatide 80 mcg SC daily for 18 months.
- Total: Total of all reporting groups
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate | Total
Number analyzed (Participants) | 558 | 581 | 1139
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 106 | 114 | 220
  65 to <74 years | 351 | 370 | 721
  ≥75 years | 101 | 97 | 198
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 558 | 581 | 1139
  Male | 0 | 0 | 0
Lumbar Spine Bone Mineral Density (BMD) T-Score [Mean (Standard Deviation); unit: T-score] — BMD data measured by a Dual Energy X-ray Absorptiometry (DXA) instrument manufactured by Lunar Prodigy or Hologic. At Baseline, participants were required to have a BMD T-score ≤2.5 to >-5.0 at the lumbar spine (L1-L4) or if the pre-specified fracture criteria were not met then T-score could be ≤3.0 to >-5.0. Osteoporosis status was based on the World Health Organization (WHO) 2007 criteria of normal (T-score >-1.0), osteopenia (T-score >-2.5 to ≤-1.0), and osteoporosis (T-score ≤-2.5). Population: All Study BA058-05-003 ITT participants who enrolled in the BA058-05-005 study (Study BA058-05-005 ITT Population) with an evaluable lumbar spine BMD T-score. Study BA058-05-003 ITT population included all participants who were randomized into the BA058-05-003 study.
  T-score
    number analyzed (Participants) | 556 | 581 | 1137
    (all) | -2.11 (0.997) | -2.87 (0.867) | -2.50 (1.008)
Femoral Neck BMD T-Score [Mean (Standard Deviation); unit: T-score] — BMD data measured by a DXA instrument manufactured by Lunar Prodigy or Hologic. At Baseline, participants were required to have a BMD T-score ≤2.5 to >-5.0 at the femoral neck or if the pre-specified fracture criteria were not met then T-score could be ≤3.0 to >-5.0. Osteoporosis status was based on the WHO 2007 criteria of normal (T-score >-1.0), osteopenia (T-score >-2.5 to ≤-1.0), and osteoporosis (T-score ≤-2.5). Population: All Study BA058-05-003 ITT participants who enrolled in the BA058-05-005 study (Study BA058-05-005 ITT Population) with an evaluable femoral neck BMD T-score. Study BA058-05-003 ITT population included all participants who were randomized into the BA058-05-003 study.
  T-score
    number analyzed (Participants) | 555 | 581 | 1136
    (all) | -1.951 (0.656) | -2.196 (0.695) | -2.077 (0.687)
Total Hip BMD T-Score [Mean (Standard Deviation); unit: T-score] — BMD data measured by a DXA instrument manufactured by Lunar Prodigy or Hologic. At Baseline, participants were required to have a BMD T-score ≤2.5 to >-5.0 at the femoral neck or if the pre-specified fracture criteria were not met then T-score could be ≤3.0 to >-5.0. Osteoporosis status was based on the WHO 2007 criteria of normal (T-score >-1.0), osteopenia (T-score >-2.5 to ≤-1.0), and osteoporosis (T-score ≤-2.5). Population: All Study BA058-05-003 ITT participants who enrolled in the BA058-05-005 study (Study BA058-05-005 ITT Population) with an evaluable femoral neck BMD T-score. Study BA058-05-003 ITT population included all participants who were randomized into the BA058-05-003 study.
  T-score
    number analyzed (Participants) | 555 | 581 | 1136
    (all) | -1.63 (0.742) | -1.93 (0.758) | -1.78 (0.765)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥1 New Vertebral Fracture Since Study BA058-05-003 Baseline
Description: Vertebral fractures were determined clinically and via protocol directed radiograph evaluation. Complete results for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Time Frame: Study BA058-05-003 Baseline (Day 1) up to Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Population: Study BA058-05-005 mITT Population: all Study BA058-05-003 mITT participants with a Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25) evaluable radiologic assessment (spine X-ray). Study BA058-05-003 mITT population included all ITT participants with a pretreatment and postbaseline evaluable radiologic assessment during Study BA058-05-003.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 544 | 568
Participants | 3 | 25

2. Secondary Outcome: Number of Participants With a Nonvertebral Fracture Since Study BA058-05-003 Baseline (Data From Studies BA058-05-005 and BA058-05-003 Combined)
Description: Nonvertebral fractures were defined as clinical fractures that included: 1) those of the hip, wrist, forearm, shoulder, collar bone, upper arm, ribs, upper leg (not hip), knee, lower leg (not knee or ankle), foot, ankle, hand, pelvis (not hip), tailbone, and other; and 2) those associated with low trauma, defined as a fall from standing height or less; a fall on stairs, steps or curbs; a minimal trauma other than a fall; or moderate trauma other than a fall. Complete results for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Time Frame: Study BA058-05-003 Baseline (Day 1) up to Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Population: Study BA058-05-005 ITT Population: all Study BA058-05-003 ITT participants who enrolled in the BA058-05-005 study. Study BA058-05-003 ITT population included all participants who were randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 558 | 581
Participants | 15 | 32

3. Secondary Outcome: Percent Change From Study BA058-05-003 Baseline in Total Hip BMD at Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Description: Total hip BMD were measured via DXA. Complete results for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Time Frame: Study BA058-05-003 Baseline (Day 1), Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Population: Study BA058-05-005 ITT Population: all Study BA058-05-003 ITT participants who enrolled in the BA058-05-005 study. Study BA058-05-003 ITT population included all participants who were randomized into Study BA058-05-003. Missing BMD data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 558 | 581
percent change | 5.4737 (3.9884) | 1.3698 (2.9712)

4. Secondary Outcome: Percent Change From Study BA058-05-003 Baseline in Femoral Neck BMD at Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Description: Femoral neck BMD were measured via DXA. Complete results for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Time Frame: Study BA058-05-003 Baseline (Day 1), Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 558 | 581
percent change | 4.5113 (4.8042) | 0.4649 (3.7913)

5. Secondary Outcome: Percent Change From Study BA058-05-003 Baseline in Lumbar Spine BMD at Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Description: Lumbar spine BMD were measured via DXA. Complete results for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Time Frame: Study BA058-05-003 Baseline (Day 1), Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 558 | 581
percent change | 12.7921 (7.9790) | 3.5133 (4.2765)

6. Secondary Outcome: Kaplan-Meier Estimated Event Rate of the First Incident of Nonvertebral Fracture Since Study BA058-05-003 Baseline (Data From Studies BA058-05-005 and BA058-05-003 Combined)
Description: as for outcome 2
Time Frame: Study BA058-05-003 Baseline (Day 1) up to Study BA058-05-005 Month 6 (Study BA058-05-003 Month 25)
Population: as for outcome 2
Measure: Number; unit: percentage of events
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 558 | 581
percentage of events | 2.7 | 5.6

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) (Data From Study BA058-05-005 Only)
Description: A TEAE is any untoward medical occurrence or undesirable event(s) experienced in a participant that begins or worsens following administration of study drug, whether or not considered related to study drug by Investigator. A serious adverse event (SAE) was an adverse event (AE) resulting in any of the following outcomes or deemed significant for any other reason, death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), congenital anomaly/birth defect, or persistent or significant disability/incapacity. Intensity for each AE was defined as mild, moderate, or severe. AEs included both SAEs and non-serious AEs. AEs whose causal relation was characterized as Possible or Probable were considered as related to study drug. AEs were coded using Medical Dictionary for Regulatory Activities (MedDRA). A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Study BA058-05-005 Baseline (Day 1) up to Study BA058-05-005 Month 24
Population: Study BA058-05-005 Safety Population: all Study BA058-05-005 ITT participants who received 1 or more doses of alendronate.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 553 | 580
Participants
  TEAEs | 452 | 466
  TEAEs Related to Study Treatment | 85 | 80
  Severe TEAEs | 38 | 40
  Serious TEAEs | 65 | 58
  TEAEs Leading to Death | 0 | 2
  TEAEs Leading to Discontinuation | 30 | 36

8. Secondary Outcome: Number of Participants With a Clinically Notable Serum Chemistry Laboratory Value (Data From Study BA058-05-005 Only)
Description: Serum Chemistry laboratory parameters that were evaluated via notable criteria (presented in parentheses) included: sodium (Low: ≤129; High: ≥148 milliequivalent per liter [mEq/L]), potassium (Low: ≤3.2; High: ≥5.5 mEq/L), albumin (<2.5 grams [g]/deciliter [dL]), total protein (<5 g/dL), glucose (Low: ≤54; High: >125 mg/dL [fasting] or >200 milligrams [mg]/dL [random]), creatinine (≥2.1 mg/dL), aspartate aminotransferase (AST) (≥5.1*upper limit of normal [ULN]), alanine aminotransferase (ALT) (≥5.1*ULN), alkaline phosphatase (AP) (≥3.1*ULN), total bilirubin (≥1.51*ULN [with any increase in liver function tests] ≥2.0*ULN [with normal liver function tests]), creatine kinase (≥3.1*ULN), total cholesterol (>226 mg/dL), and total calcium (Low: ≤7.4; High: ≥11.6 mg/dL). Only the serum chemistry parameters with at least 1 participant with a notable laboratory value are presented.
Time Frame: Study BA058-05-005 Baseline (Day 1) up to Study BA058-05-005 Month 24
Population: All Study BA058-05-005 ITT participants who received 1 or more doses of alendronate (Study BA058-05-005 Safety Population) with available data for the respective serum chemistry parameter. Only participants with a notable laboratory value are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 553 | 580
Participants
  Alkaline Phosphatase: number analyzed (Participants) | 545 | 580
  Alkaline Phosphatase | 1 | 0
  Cholesterol Total: number analyzed (Participants) | 342 | 358
  Cholesterol Total | 75 | 73
  Creatine Kinase: number analyzed (Participants) | 545 | 568
  Creatine Kinase | 2 | 1
  Glucose (Fasting; High): number analyzed (Participants) | 515 | 543
  Glucose (Fasting; High) | 22 | 18
  Glucose (Random): number analyzed (Participants) | 515 | 543
  Glucose (Random) | 1 | 2
  Potassium (Low): number analyzed (Participants) | 541 | 565
  Potassium (Low) | 1 | 3
  Potassium (High): number analyzed (Participants) | 541 | 565
  Potassium (High) | 4 | 3
  Sodium (Low): number analyzed (Participants) | 542 | 570
  Sodium (Low) | 1 | 1
  Sodium (High): number analyzed (Participants) | 542 | 580
  Sodium (High) | 6 | 2

9. Secondary Outcome: Number of Participants With a Clinically Notable Hematology Laboratory Value (Data From Study BA058-05-005 Only)
Description: Hematology laboratory parameters that were evaluated via notable criteria (presented in parentheses) included: Absolute Eosinophils (>5000 cells/mm^3), Absolute Lymphocytes (≤499 cells/mm^3), Absolute Neutrophils (≤999 cells/mm^3), % Eosinophils (>50%), % Lymphocytes (≤5%), % Neutrophils (≤10%), Hemoglobin (Low: ≤9.4 g/dL; High: change from baseline ≥2.1 g/dL), Platelets (≤99000 cells/mm^3), and White Blood Cells (Low: ≤1499 cells/mm^3; High: ≥20001 cells/mm^3). Only the hematology parameters with at least 1 participant with a notable laboratory value are presented.
Time Frame: Study BA058-05-005 Baseline (Day 1) up to Study BA058-05-005 Month 24
Population: All Study BA058-05-005 ITT participants who received 1 or more doses of alendronate (Study BA058-05-005 Safety Population) with available data for the respective hematology parameter. Only participants with a notable laboratory value are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 553 | 580
Participants
  Absolute Lymphocytes: number analyzed (Participants) | 380 | 392
  Absolute Lymphocytes | 15 | 11
  Lymphocytes (Absolute Count or Percentage): number analyzed (Participants) | 521 | 540
  Lymphocytes (Absolute Count or Percentage) | 15 | 11
  Absolute Neutrophils: number analyzed (Participants) | 392 | 410
  Absolute Neutrophils | 0 | 2
  Neutrophils (Absolute Count or Percentage): number analyzed (Participants) | 533 | 558
  Neutrophils (Absolute Count or Percentage) | 0 | 2
  Hemoglobin (Low): number analyzed (Participants) | 544 | 580
  Hemoglobin (Low) | 7 | 2
  Hemoglobin (High): number analyzed (Participants) | 544 | 580
  Hemoglobin (High) | 19 | 17
  Platelets: number analyzed (Participants) | 545 | 565
  Platelets | 1 | 0

10. Secondary Outcome: Number of Participants With a Clinically Notable Coagulation Laboratory Value (Data From Study BA058-05-005 Only)
Description: Coagulation laboratory parameters that were evaluated via notable criteria (presented in parentheses) included: Activated Partial Thromboplastin Time (≥1.41*ULN), Prothrombin Time (≥1.21*ULN). Because the Activated Partial Thromboplastin Time was the only coagulation laboratory parameter with at least 1 participant with a notable laboratory value, this is the only parameter presented below.
Time Frame: Study BA058-05-005 Baseline (Day 1) up to Study BA058-05-005 Month 24
Population: All Study BA058-05-005 ITT participants who received 1 or more doses of alendronate (Study BA058-05-005 Safety Population) with available data for the respective coagulation parameter. Only participants with a notable laboratory value are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 553 | 580
Participants | 9 | 4

11. Secondary Outcome: Number of Participants With a Clinically Notable Urine Laboratory Value (Data From Study BA058-05-005 Only)
Description: Urine laboratory parameters that were evaluated via notable criteria (presented in parentheses) included: Glucose (2+), Protein (2+), Blood (>50 red blood cells per high-power field [rbc/hpf]).
Time Frame: Study BA058-05-005 Baseline (Day 1) up to Study BA058-05-005 Month 24
Population: All Study BA058-05-005 ITT participants who received 1 or more doses of alendronate (Study BA058-05-005 Safety Population) with available data for the respective urine laboratory parameter. Only participants with a notable laboratory value are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Number analyzed (Participants) | 553 | 580
Participants
  Glucose | 4 | 3
  Protein: number analyzed (Participants) | 543 | 567
  Protein | 6 | 6
  Blood: number analyzed (Participants) | 482 | 496
  Blood | 77 | 50

ADVERSE EVENTS:
Time Frame: Study BA058-05-005 Baseline (Day 1) up to Study BA058-05-005 Month 24
Description: Study BA058-05-005 Safety Population: all Study BA058-05-005 ITT participants who received 1 or more doses of alendronate. Serious and Non-Serious TEAEs are presented. Adverse events for Study BA058-05-003 are reported in the ClinicalTrials.gov Study Record NCT02653417.
Arm/Group | Abaloparatide-SC/Alendronate | Placebo/Alendronate
Serious Adverse Events (participants affected / at risk) | 65/553 | 58/580
Other Adverse Events (participants affected / at risk) | 145/553 | 158/580
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide-SC/Alendronate (N=553) | Placebo/Alendronate (N=580)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 1
Retinal detachment (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Drug induced liver injury (Hepatobiliary disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 1
Pericarditis infective (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Viral myositis (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 3
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebellar ischaemia (Nervous system disorders) | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 4 | 0
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Medical device removal (Surgical and medical procedures) | 0 | 1
Nasal septal operation (Surgical and medical procedures) | 1 | 0
Removal of internal fixation (Surgical and medical procedures) | 1 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide-SC/Alendronate (N=553) | Placebo/Alendronate (N=580)
Upper respiratory tract infection (Infections and infestations) | 40 | 51
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 | 58
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 34
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 31
Hypertension (Vascular disorders) | 27 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes